CLINICAL TRIAL: NCT00673764
Title: The Effect of Systane Ultra Lubricant Eye Drops (FID 112903) on Visual Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-07-24
Record Dates: First submitted 2008-05-02; First posted 2008-05-07 (Estimated); Results first posted 2010-02-10 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane Ultra (Experimental): Systane Ultra Lubricant Eye Drops
  Interventions: Other: Systane Ultra Lubricant Eye Drops
- Optive (Active Comparator): Optive Lubricant Eye Drops
  Interventions: Other: Optive Lubricant Eye Drops

INTERVENTIONS:
Other: Systane Ultra Lubricant Eye Drops — Systane Ultra Lubricant Eye Drops 1 drop each eye one time
  Arms: Systane Ultra
Other: Optive Lubricant Eye Drops — Optive Lubricant Eye Drops 1 drop each eye one time
  Arms: Optive

SUMMARY:
To evaluate the effect of 2 different lubricant eye drops on visual function of patients with dry eye

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of dry eye
* Must not have worn contact lenses for 12 hours prior to Day 1

Exclusion Criteria:

* Age related

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- North Andover, North Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 48 Dry Eye Subjects
Pre-assignment Details: Randomized, double-masked, crossover
Groups:
- Systane Ultra, Then Optive: Systane Ultra Lubricant Eye Drops first, then cross-over to Optive.
- Optive, Then Systane Ultra: Optive Lubricant Eye Drops first, then cross-over to Systane Ultra.
Period: Overall Study
Arm/Group | Systane Ultra, Then Optive | Optive, Then Systane Ultra
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Overall Study
Arm/Group | Overall Study
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Time at Best Corrected Visual Acuity
Description: Measuring length of time patient can maintain their best vision while completing a computer task. Performed at 15 minutes, 45 minutes, and 90 minutes post-dose. Corrected visual acuity means the patient can wear glasses or contacts if needed such that the measure is performed with the patient seeing the best that they can.
Time Frame: 15 minutes, 45 minutes, and 90 minutes post-dose
Measure: Median (Standard Error); unit: seconds
Arm/Group | Systane Ultra | Optive
Number analyzed (Participants) | 48 | 48
seconds
  15 minutes post-dose | 7.75 (0.6545) | 6.42 (.6545)
  45 minutes post-dose | 6.46 (0.4003) | 5.51 (0.4003)
  90 minutes post-dose | 9.17 (0.0365) | 6.84 (0.0365)

2. Secondary Outcome: Functional Blink Rate Time (Time Between Blinks)
Description: Measures time in seconds between normal blinks. Performed at 15 minutes, 45 minutes, and 90 minutes post-dose. Longer blink rate time correlates with improved visual performance.
Time Frame: 15 minutes, 45 minutes, and 90 minutes post-dose
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Systane Ultra | Optive
Number analyzed (Participants) | 48 | 48
seconds
  15 minutes post-dose | 5.9 (5.5) | 5.8 (4.7)
  45 minutes post-dose | 5.9 (5.4) | 6.7 (4.9)
  90 minutes post-dose | 6.5 (5.8) | 7.3 (6.0)

ADVERSE EVENTS:
Arm/Group | Systane Ultra | Optive
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI should hold confidential, and not disclose directly or indirectly to any third party other than Contractors, the data arising out of the study. Alcon reserves the right of prior review of any publication or presentation of information related to the study.